CLINICAL TRIAL: NCT02602236
Title: Multicenter Pilot Study to Describe the Performance of a New Device in Patients With Colostomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigational product needs improvements
Sponsor: BBraun Medical SAS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OPM-G-H-1401; 2015-A00611-48 (Other: FRENCH HEALTH AUTORITY)
Record Dates: First submitted 2015-11-04; First posted 2015-11-11 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Colostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AOS-C2000-B (Experimental): A new 2-piece appliance composed with 2 parts : a base plate and an ostomy collection special pouch (1 base plate for 2 or 3 days and 1 to 4 collection special pouch per day)
  Interventions: Device: AOS-C2000-B

INTERVENTIONS:
Device: AOS-C2000-B — 1 base plate for 2 or 3 days and 1 to 4 collection special pouch per day

SUMMARY:
The study evaluates the efficacy of a new 2-piece appliance in patients with colostomy.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years old
* Patient having a colostomy with a diameter less than 30 mm for users of Ø 55 mm pouches or having a colostomy with a diameter less than 40 mm for users of Ø 65 mm pouches
* Patient having a colostomy for at least 1 month
* Patient using currently the two-piece flat ostomy appliance Flexima®/Softima® 3S for at least 2 weeks and being satisfied
* Patient having a stoma protusion smaller than or equal to 1.5 cm
* Patient capable to apply and remove the appliance himself or with the help of a caregiver (except health care professional)
* Patient having a mental capacity to participate to the study (i.e. to understand the study and to answer to the questions)
* Patient agreeing to test the new appliance during the training phase (5±3 days) and during the study device usage phase (14±3 days)
* Patient covered by social security

Exclusion Criteria:

* Patient experiencing repeated leakages with the usual pouching system
* Patient currently suffering from peristomal skin complications (bleeding or red and broken skin at the time of inclusion)
* Patient receiving or having received, within the last month, chemotherapy, radiotherapy or corticotherapy
* Patient already participating in another clinical study or who have previously participated in this investigation
* Pregnant or breast-feeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-11; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Description of efficacy in term of type of bag deployment and leakage prevention | At least 1 time per day during 14±3 days
  After each change of the investigational product, the patient will describe on a 3-point scale the type of deployment "manual", "spontaneous - in link with stools or gas", "spontaneous - no link with stools or gas"

SECONDARY OUTCOMES:
Peristomal skin evaluation with DET score scale | baseline and 5±3 days and 14±3 days
Investigational product bag deployment reason | At each bag change during 14±3 days
  Evaluation with a questionnaire (4-points very satisfying to not at all satisfying)
Ease of bag deployment | 14±3 days
  Evaluation with a questionnaire (4-points very satisfying to not at all satisfying)
Ease of special bag handling | 14±3 days
  Evaluation with a questionnaire (4-points very satisfying to not at all satisfying)
Investigational product bag ease of use of gas release button | 14±3 days
  Evaluation with a questionnaire (4-points very satisfying to not at all satisfying)
Ease of control of gas release button | 14±3 days
  Evaluation with a questionnaire (4-points very satisfying to not at all satisfying)
General impression about the investigational device before use | 14±3 days
  Evaluation with a questionnaire (4-points very satisfying to not at all satisfying)
Investigational device wearing comfort | 14±3 days
  Evaluation with a questionnaire (4-points very satisfying to not at all satisfying)
Investigational device flexibility | 14±3 days
  Evaluation with a questionnaire (4-points very satisfying to not at all satisfying)
Investigational device discretion | 14±3 days
  Evaluation with a questionnaire (4-points very satisfying to not at all satisfying)
Ease of base plate handling | 14±3 days
  Evaluation with a questionnaire (4-points very satisfying to not at all satisfying)
Investigational device adhesivity during wear time | 14±3 days
  Evaluation with a questionnaire (4-points very satisfying to not at all satisfying)
Investigational device filter performance with deployed bag | 14±3 days
  Evaluation with a questionnaire (4-points very satisfying to not at all satisfying)
Investigational device filter performance with undeployed bag | 14±3 days
  Evaluation with a questionnaire (4-points very satisfying to not at all satisfying)
Efficacy of Investigational device gas release button | 14±3 days
  Evaluation with a questionnaire (4-points very satisfying to not at all satisfying)
Noise during Investigational device wear time | 14±3 days
  Evaluation with a questionnaire (4-points very satisfying to not at all satisfying)
Overall satisfaction questionnaire of the collection volume of the bag of the Investigational device | 14±3 days
Overall security feeling questionnaire with the Investigational device | 14±3 days
Overall satisfaction questionnaire with the Investigational device | 14±3 days
Overall satisfaction questionnaire regarding bag deployment of the Investigational device | 14±3 days
Overall satisfaction questionnaire with cap cover of the Investigational device | 14±3 days
General impression about body image during use of the investigational product | 14±3 days
  (4-points very satisfying to not at all satisfying)
Assessment questionnaire of willingness to use and the frequency of use in the future | 14±3 days
Assessment of the investigational device wear time | 14±3 days
Assessment questionnaire preference between the investigational device and usual appliance | 14±3 days
Assessment of use of accessories | At each bag change during 14±3 days
  Choice between some accessories
Assessment of the quality of life with Stoma-QoL questionnaire | At baseline, at 5±3 days and 14±3 days
Number of participants with Adverse Event as a measure of safety and tolerability | At baseline, at 5±3 days and 14±3 days

CONTACTS AND LOCATIONS:
Overall Officials: Mahaut LECONTE, MD, Principal Investigator — University Hospital of Paris - Cochin
Locations (1):
- Centre Georges François Leclerc, Dijon, France